CLINICAL TRIAL: NCT00301197
Title: Childhood Obesity Treatment: A Maintenance Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5R01HD036904 (NIH)
Record Dates: First submitted 2006-03-08; First posted 2006-03-10 (Estimated); Last update posted 2006-03-10 (Estimated); Status verified 2006-03

CONDITIONS: Obesity
Keywords: Childhood obesity; intervention; obesity; weight loss; behavior therapy; peer group; social support network; child; clinical research; human subject
MeSH Terms: conditions — Obesity; Pediatric Obesity; Weight Loss

INTERVENTIONS:
Behavioral: Behavioral Skills Maintenance
Behavioral: Social Facilitation Maintenance

SUMMARY:
Obesity is a major public health problem. At least 15 million American adults are obese, and the number is rising. Childhood obesity is also increasing in prevalence and currently affects approximately 11-22 percent of children aged 6 to 11. Childhood obesity is associated with serious negative physical, emotional, and social consequences. Obese children are at high risk for becoming obese as adults; 24-44 percent of obese adults were obese as children. The risk of an obese child becoming an obese adult is especially high when at least one parent is obese. To date, adult obesity is known to be resistant to treatment. In contrast, promising long-term effects have been found with children who received behavioral family-based weight loss treatment. However, even with state-of-the-science programs, a substantial percentage of children (i.e., over 40 percent) regain all or most of the weight lost once treatment ends. The proposed study examined the efficacy of two intervention strategies designed to improve the long-term maintenance of weight loss in children relative to discontinued treatment contact following an active weight loss treatment phase (no maintenance treatment control (NTC).

DETAILED DESCRIPTION:
This is an efficacy study comparing two intervention strategies designed to improve the long-term maintenance of weight loss in children compared to a no maintenance treatment control group. In this study, overweight children between the ages of 7-12 years old participated along with their overweight parents in a 20-week behavioral, family-based weight loss treatment. Following weight loss treatment, participants were randomly assigned to one of two 4-month maintenance interventions or to a no-continued treatment control. The Behavioral Skills Maintenance intervention (BSM) will confront the declining motivation to engage in weight-maintenance behaviors, incorporate specific skills for weight maintenance, and teach coping skills and relapse prevention techniques. The Social Facilitation Maintenance treatment will use an innovative, socially-based approach to enhance peer support, increase parental instrumental support, improve body image, and teach effective responses to teasing as methods for sustaining weight maintenance behaviors (i.e., healthy diet and physical activity). It is expected that children participating in BSM and SFM interventions will demonstrate better outcomes at the point of the weight maintenance intervention cessation than children not provided any maintenance treatment. It is further hypothesized that the developmentally appropriate focus and more pervasive and sustaining nature of the SFM treatment targets relative to BSM targets will result in better weight maintenance outcomes for SFM than BSM children. Follow-up assessments will occur at the end of the maintenance phase of treatment, as well as at 12 and 24 months following the initial weight loss treatment. Effective maintenance treatments in children will have a substantial impact on children's immediate and future physical, psychological, and social well being.

ELIGIBILITY:
Inclusion Criteria:

Child:

* 20%-100% overweight
* 7-12 years old

At least one parent:

* At least 20% overweight
* Actively participates in program along with participating child

Both participating family members:

* Can read and speak English at a 3rd grade level

Exclusion Criteria:

Either participating child or parent:

* has current psychopathology and is not in ongoing psychiatric care
* has an active substance abuse problem
* is not taking weight-affecting medications
* does not have a medical condition for which a weight loss program would be contraindicated
* does not have a physical disability of illness that limits their ability to do physical activity
* does not have major dietary restrictions
* is not participating in an active weight loss treatment

All family members:

* do not have an active eating disorder

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 216
Dates: Start 1999-08; Study Completion 2004-04

PRIMARY OUTCOMES:
Weight (child and parent)

SECONDARY OUTCOMES:
Weight related behaviors
Psychological functioning (specific and general)

CONTACTS AND LOCATIONS:
Overall Officials: Denise E Wilfley, PhD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- [Derived] Wilfley DE, Stein RI, Saelens BE, Mockus DS, Matt GE, Hayden-Wade HA, Welch RR, Schechtman KB, Thompson PA, Epstein LH. Efficacy of maintenance treatment approaches for childhood overweight: a randomized controlled trial. JAMA. 2007 Oct 10;298(14):1661-73. doi: 10.1001/jama.298.14.1661. PMID 17925518